CLINICAL TRIAL: NCT05311722
Title: Comparing the Efficacy of Intravenous Dexmedetomidine, Tramadol and Ketamine for Control of Post Spinal Shivering in Obstetric Patients Undergoing Lower Segment C-section
Brief Title: Comparsion of IV Dexmedetomidine, Tramdol and Ketamine for Post Spinal Anesthesia Shivering.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheikh Zayed Medical College (Other Government)
Responsible Party: Principal Investigator, Obaid ur Rehman, Principal investigator, Sheikh Zayed Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ORehman
Record Dates: First submitted 2022-03-09; First posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Post-Surgical Complication
MeSH Terms: interventions — Dexmedetomidine; Ketamine; Tramadol

STUDY DESIGN:
Intervention Model Description: 3 drugs were given to patients
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dexmedetomidine (Experimental): Inj.dexmedetomidine 0.5mcg/kg diluted in 10ml N/s given as iv infusion over 10 minutes
  Interventions: Drug: Dexmedetomidine
- Ketamine (Experimental): Inj.ketamine 0.5mg/kg diluted in 10ml N/s given as iv infusion over 10 minutes
  Interventions: Drug: Ketamine
- Tramadol (Experimental): Inj.tramadol 0.5mg/kg diluted in 10ml N/s given as iv infusion over 10 minutes
  Interventions: Drug: Tramadol

INTERVENTIONS:
Drug: Dexmedetomidine — Inj dexmedetomidine, will be given in infusion over 10 mins and their effect on post spinal shivering will be assessed.
  Arms: Dexmedetomidine
Drug: Ketamine — Ketamine
  Arms: Ketamine
Drug: Tramadol — Tramadol
  Arms: Tramadol

SUMMARY:
To study control of post spinal shivering in patients undergoing lower segment cesarean section using dexmedetomidine, tramadol and ketamine

DETAILED DESCRIPTION:
Its a Comparison of drugs for a better control of post spinal shivering in patietns underwent cesarean section.using grades of shivering (0-4)patients will be assessed

ELIGIBILITY:
Inclusion Criteria:

* Woman of age 18-60
* Pregnant woman in outdoor patient department and emergency

Exclusion Criteria:

* patient. with history of hypersensitivity to opioids,
* ketamine or bupivacaine
* History of cardiovascular disease,
* Hypertension,
* psychosis,
* antepartum hemorrhage,
* cord prolapse,
* fetal distress

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — All females with age between 18 -60
Enrollment: 71 (Estimated)
Dates: Start 2022-04-30 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-02-20 (Estimated)

PRIMARY OUTCOMES:
Assessment of post spinal shivering by observing grades of shivering | 10 minutes
  Control of post spinal shivering dexmedetomidine, tramadol and ketamine for control of post spinal shivering.

IPD SHARING:
Plan to Share IPD: No